CLINICAL TRIAL: NCT04107233
Title: Using Electronic Medical Record Data to Improve HIV Primary Care: an Audit and Feedback Study
Brief Title: Using Electronic Medical Record Data to Improve HIV Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SMH-16-381
Record Dates: First submitted 2019-05-31; First posted 2019-09-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Quality of Health Care; HIV/AIDS; Electronic Health Records
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Audit and feedback directed at family physicians, including reports a one-on-one meeting.
  Interventions: Behavioral: Audit and Feedback
- Control (No Intervention): Usual care; may receive the intervention at the end of the study if successful

INTERVENTIONS:
Behavioral: Audit and Feedback — Charts for enrolled physicians will be audited and they will receive feedback, consisting of tailored reports and one-on-one meeting with colleague to review at baseline, 3 months and 6 months
  Arms: Intervention

SUMMARY:
This cluster randomized control trial examines whether an audit and feedback study improves care of patients living with HIV/AIDS in a family health team setting.

DETAILED DESCRIPTION:
This cluster randomized control trial will use electronic medical record (EMR) data from the St. Michael's Hospital Academic Family Health Team to examine whether the quality of HIV care provided to patients can be improved through an audit and feedback (A&F) intervention. Our objective is to examine whether A&F targeting family physicians caring for people living with HIV/AIDS (PHLA) using EMR data can improve laboratory monitoring, engagement in primary care and the uptake of preventive interventions.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians at the St. Michael's Hospital Academic Family Health Team who have at least 20 PLHA.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Up to date viral load | Within six months
  Percentage of HIV infected patients who have an up to date HIV viral load

SECONDARY OUTCOMES:
Clinic visit | Within the last 6 months
  To assess engagement in care (number of patients who went to see a physician)
Up-to-date cancer screenings | 1-3 years
  Presence of cancer monitoring for colorectal, breast and cervical cancers
Vaccinations | Since 2013
  Up-to-date for both pneumococcal vaccines and seasonal influenza vaccine (number of patients who received a specific vaccination)
Screening for diabetes | Within 1 year
  For those 40 or older, the presence of either a fasting blood glucose or HbA1c in the chart
Screening for hypercholesterolemia | Within 1 year
  For those 40 or older. the presence of an LDL or non-HDL in the chart
Screening for osteoporosis | Within 5 years
  For patients 50 years and older, the presence of a bone mineral density report

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pinto, MSc MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided